CLINICAL TRIAL: NCT02404662
Title: Single Blind Randomised Trial of Supportive Text Messages for Patients With Alcohol Use Disorder and a Co-morbid Depression
Brief Title: Trial of Supportive Text Messages for Patients With Alcohol Use Disorder and a Co-morbid Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St Patrick's Hospital, Ireland (Other)
Collaborators: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Dr. Conor Farren, Associate Clinical Professor, Trinity College Dublin; Consultant Psychiatrist, St Patrick's University Hospital, St Patrick's Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HRA-POR-2014-598
Record Dates: First submitted 2015-03-19; First posted 2015-03-31 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-05

CONDITIONS: Dual Diagnosis
Keywords: Alcohol use disorder; Depression; Mood disorders; Bipolar disorder; Supportive text messages
MeSH Terms: conditions — Alcoholism; Depression; Mood Disorders; Bipolar Disorder | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supportive text messages intervention (Experimental): Patients in the intervention group will receive twice daily supportive text messages to their mobile phone for 6 months following discharge from a 4-week in-patient dual diagnosis treatment programme. The messages will be sent by a computer programme at 10am and 7pm each day and will be set up and monitored by the research worker who will not participate in follow-up assessments. They will receive a fortnightly text message thanking them for participating in the study, and a brief phone call every 2 weeks to ensure that they are still using their phone and that they have received some messages. The intervention group will also receive treatment as usual, i.e. any follow-up after-care that they chose to participate in and regular AA/Lifering meetings.
  Interventions: Other: Supportive text messages intervention
- Control group (Active Comparator): Patients in the control group will receive a fortnightly text message thanking them for participating in the study, and a brief phone call every 2 weeks to ensure that they are still using their phone and that they have received some messages. The control group will also receive treatment as usual, i.e. any follow-up after-care that they chose to participate in and regular AA/Lifering meetings.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Supportive text messages intervention — The supportive text messages are based on existing aphorisms in the recovery literature. Each day patients will receive one message targeting mood and another message targeting abstinence from alcohol in accordance with the primary aims of our study. An example text message aimed at improving mood is: "Monitor changes in your mood; develop a list of personal warning signs." An example message targeting abstinence is: "Keep Sobriety as a number one priority and you will reach your goals. None of the messages will be repeated. The messages will be sent in the morning and evening, with the theme (mood/alcohol) of the messages pseudo-randomised according to delivery time, so that no more than three successive days will have the same theme sent at the same time slot.
  Arms: Supportive text messages intervention
Other: Control group — The control group will receive treatment as usual, as well as fortnightly thank you text messages and calls to ensure that they are still using their phone.
  Arms: Control group

SUMMARY:
Most patients who present with problem drinking also present with mood problems. Problem drinking and mood problems co-occurring together in individuals lead them to have more severe symptoms, greater disability and poorer quality of life than individuals with only problem drinking, and they pose a greater economic burden to society due to their higher use of health services. This study aims to assess the efficacy of a new, innovative and cost effective treatment strategy aimed at reducing the burden that these co-occurring conditions impose on the suffers and their families as well as the community and health systems.

In a recent pilot study of supportive text messages for patients with problem drinking and co-occurring depression, the investigators established that patients who received twice daily supportive text messages for three months had significantly less depressive symptoms than those who did not receive such messages. There was also a trend to finding that patients who received the supportive text messages were more likely to have higher alcohol free days than those who did not receive any supportive text messages.

This study seeks to extend the knowledge gained from the pilot study. A larger group of patients with alcohol use disorder and a depressive disorder will be randomly assigned to two groups. One group will receive supportive text messages for six months duration whilst the other group will receive no supportive text messages. The patients will be followed up at 3, 6, 9 and 12 months to determine which of the two groups have less alcohol and mood problems. It is anticipated that patients receiving supportive text messages will report significantly greater alcohol free days as well as significantly less relapses, hospitalizations and mood symptoms than those not receiving such messages.

DETAILED DESCRIPTION:
Co-morbidity of alcohol use disorder (AUD) and mood disorders presents a great challenge to health systems and exacts a tremendous toll world-wide. Individuals with a dual diagnosis have more severe symptoms, greater disability and poor quality of life than those with either diagnosis alone, and pose a greater economic burden to society due to their higher use of treatment services. New, enhanced, efficient, innovative and cost effective treatment strategies aimed at reducing the burden that the disorders impose on the suffers and their families as well as the community and health systems are required. In a pilot trial of supportive text messages for patients with alcohol use disorders and co-morbid depression, the investigators established that patients who received twice daily supportive text messages for three months had significantly less depressive symptoms than those who did not receive such messages. There was also a trend to finding that patients who received the supportive text messages were more likely to have higher cumulative abstinence duration than those who did not receive any supportive text messages.

This research seeks to extend the knowledge gained from the pilot trial. A randomised trial will be conducted on a larger sample size of patients with alcohol use disorder and a co-morbid depressive disorder (including bipolar depression) for an extended duration (6 months of supportive text messages and 1 year follow-up instead of 3 months text messages with 6 months follow-up in the pilot trial). It is hypothesised that patients receiving supportive text messages will report significantly greater cumulative abstinence duration as well as significantly less relapses, hospitalizations and mood symptoms than those not receiving such messages. It is anticipated that this technology intervention for relapse prevention will be acceptable to patients as well as cost effective.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the criteria for both alcohol dependency syndrome/alcohol abuse and either major depressive disorder or bipolar disorder according to the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID) and are enrolled on the in-patient dual diagnosis or addiction treatment programmes in St. Patrick's University Hospital.
2. Able to provide written, informed consent.
3. Mini-mental state examination (MMSE) score of ≥ 25
4. Patients who have a mobile phone, are familiar with SMS text messaging technology and are willing to take part in the study.

Exclusion Criteria:

1. Patients who do not consent to take part in the study.
2. Patients who do not have a mobile phone or are unable to use the mobile text message technology.
3. Patients who would be unavailable for follow-up during the study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative abstinence duration (CAD). | 12 months following discharge from the inpatient treatment programme.
  CAD will be assessed using the timeline to follow-back (TLFB). This will be used to record the quantity of alcohol consumed and number of drinking days.
Changes in Beck's Depression Inventory (BDI) scores from baseline. | BDI will be administered at baseline (during the in-patient treatment programme for dual diagnosis), and then at 3, 6, 9 and 12 months post-discharge from hospital.
  The BDI is a self-administered questionnaire widely used to assess depressive symptoms. It takes approximately 5 minutes to complete.

SECONDARY OUTCOMES:
Proportion of patients continuously abstinent from alcohol at 6 and 12 months. | 6 and 12 months post-discharge.
  Continuous abstinence will be assessed using the TLFB.
Time to first drink. | 3, 6, 9 and 12 months post-discharge.
  The time between the patient's discharge from hospital and their first drink, if any, during the study, will be measured using the TLFB.
Perception of patients in the intervention group about the usefulness of supportive text messages. | 6 months post-discharge
  Patient perceptions about the usefulness of the intervention will be assessed at the end of the intervention period in an interview.
Changes from baseline in scores on the modified global assessment of function (m-GAF) scale. | This assessment will be completed at baseline and then at 3, 6, 9 and 12 months.
  The m-GAF will be used to measure subjective changes in the social, occupational and psychological functioning of the patients over the course of the study.
Changes from baseline in scores on the alcohol expectancy questionnaire (AEQ). | This scale will be administered at baseline and then at 3, 6, 9 and 12 months.
  This scale will measure changes in attitudes towards alcohol over the course of the study.
Changes from baseline in scores on the obsessive compulsive drinking scale (OCDS). | This scale will be administered at baseline and then at 3, 6, 9 and 12 months.
  This scale will measure changes in obsessive compulsive thoughts about alcohol over the 12 months of the study.
Changes from baseline in scores on the alcohol abstinence self-efficacy scale (AASES). | These scales will be administered at baseline and then at 3, 6, 9 and 12 months.
  This scale will measure changes in feelings of self-efficacy and personal control around drinking over the 12 months of the study.
Changes from baseline in scores on the perceived stress scale (PSS). | This scale will be administered at baseline and then at 3, 6, 9 and 12 months.
  This scale will measure changes in perceived stress over the 12 months of the study. This construct is closely related to resilience, which is a positive predictor of recovery in addiction.
Changes from baseline in scores on the young mania rating scale (YMRS). | This assessment will be completed at baseline and then at 3, 6, 9 and 12 months.
  This subjective rating scale assesses the level of mania in patients with bipolar disorder (BP). It will be used to track changes in the manic symptoms of the BP patients over the 12 months of the study.
Changes from baseline in blood measures of alcohol abuse. | Blood samples will be analysed at baseline, then at 3, 6, 9 and 12 months following discharge.
  Three blood measures suggestive of alcohol abuse will be taken to corroborate self-report measures of alcohol intake or abstinence from the TLFB- gamma glutamyl transferase (GGT), alkaline phosphatase (AST) and mean corpuscular volume (MCV).
Patient satisfaction with overall treatment protocol in both groups | 3, 6, 9 and 12 months
  Patient satisfaction will be assessed using an adaptation of a treatment evaluation questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Conor Farren, PhD,MRCPsych, Principal Investigator — St Patrick's Hospital, Ireland
Locations (1):
- St. Patrick's University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agyapong VI, Ahern S, McLoughlin DM, Farren CK. Supportive text messaging for depression and comorbid alcohol use disorder: single-blind randomised trial. J Affect Disord. 2012 Dec 10;141(2-3):168-76. doi: 10.1016/j.jad.2012.02.040. Epub 2012 Mar 29. PMID 22464008
- [Background] Agyapong VI, McLoughlin DM, Farren CK. Six-months outcomes of a randomised trial of supportive text messaging for depression and comorbid alcohol use disorder. J Affect Disord. 2013 Oct;151(1):100-4. doi: 10.1016/j.jad.2013.05.058. Epub 2013 Jun 22. PMID 23800443
- [Background] Agyapong VI, Milnes J, McLoughlin DM, Farren CK. Perception of patients with alcohol use disorder and comorbid depression about the usefulness of supportive text messages. Technol Health Care. 2013;21(1):31-9. doi: 10.3233/THC-120707. PMID 23358057
- [Derived] Hartnett D, Murphy E, Kehoe E, Agyapong V, McLoughlin DM, Farren C. Supportive text messages for patients with alcohol use disorder and a comorbid depression: a protocol for a single-blind randomised controlled aftercare trial. BMJ Open. 2017 May 29;7(5):e013587. doi: 10.1136/bmjopen-2016-013587. PMID 28554910